CLINICAL TRIAL: NCT00622076
Title: Randomised Controled Multicenter Trial Regarding the Appropriate Length of Postoperative Catheterization After Anterior Colporrhaphy for Repair of Cystocele
Brief Title: Postoperative Catheterization After Anterior Colporrhaphy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atrium Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Weemhoff, Atrium medical center Heerlen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-P-47
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-01

CONDITIONS: Cystocele; Cystitis
Keywords: postoperative; Catheterization; colporrhaphy; cystocele; cystitis
MeSH Terms: conditions — Cystocele; Cystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): postoperative catheterization after anterior colporrhaphy during five days.
  Interventions: Procedure: postoperative catheterization
- 2. (Active Comparator): postoperative catheterization after anterior colporrhaphy during two days
  Interventions: Procedure: postoperative catheterization

INTERVENTIONS:
Procedure: postoperative catheterization — postoperative catheterization after anterior colporrhaphy for five days versus two days.
  Other Names: catheterization protocol

SUMMARY:
Randomised controled multicenter trial about the appropriate length of postoperative catheterization after anterior colporrhaphy. Patients are included at the moment that they are planned for surgery and are allocated to one of the study arms after the operation in the recovery by a digital randomisation-procedure. 230 patients will be enrolled in the study and half of the patients will have a catheter during five days postoperatively and the other half will be catheterized only during two days. Main outcome measurements regards replacement of a catheter because of bladder retention and the occurence of cystitis.

ELIGIBILITY:
Inclusion Criteria:

* all patients planned for a cystocele repair

Exclusion Criteria:

* patients who already have voiding problems before the operation not related to the cystocele
* patients that are not capable of understanding our patient information form because of mental status or language

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
how many patients do need replacement of a catheter because of urine retention in both groups: 2 days versus 5 days in dwelling catheterization after anterior colporrhaphy | 6-8 hours after removal of catheter

SECONDARY OUTCOMES:
how many patients develop cystitis after catheterization in both groups: 2 days versus 5 days in dwelling catheterization after anterior colporrhaphy | 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frans Roumen, Dr, Study Director — Atrium Medical Center; Mirjam Weemhoff, DRS, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - atriumMC, Heerlen
  - Maastricht university medical center, Maastricht

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246